CLINICAL TRIAL: NCT01032083
Title: Individually Randomised, Placebo-controlled, Parallel Arm RCT With 12-month Follow-up to Establish the Clinical and Cost Effectiveness of the Antidepressant Citalopram in the Management of Negative Symptoms of Schizophrenia
Brief Title: Antidepressant Controlled Trial for Negative Symptoms in Schizophrenia
Acronym: ACTIONS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Manchester (Other); University of Southampton (Other); King's College London (Other); University of Oxford (Other); University College, London (Other); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO 1250; 2009-009235-30 (EudraCT Number)
Record Dates: First submitted 2009-08-04; First posted 2009-12-15 (Estimated); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia
Keywords: SSRI antidepressant; Negative symptoms; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram (Active Comparator): An SSRI antidepressant
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — Treatment with citalopram will be initiated at 20mg/day for the first 4 weeks (or one placebo capsule), followed by the option to increase the dose to 40mg per day (or two placebo capsules) for the remainder of the study period.
  Arms: Citalopram
Drug: Placebo — Treatment with citalopram will be initiated at 20mg/day for the first 4 weeks (or one placebo capsule), followed by the option to increase the dose to 40mg per day (or two placebo capsules) for the remainder of the study period.
  Arms: Placebo

SUMMARY:
The aim of this double-blind, placebo-controlled trial is to establish the clinical and cost effectiveness of an SSRI antidepressant, citalopram, in the management of persistent negative symptoms of schizophrenia over a year.

DETAILED DESCRIPTION:
The negative symptoms of schizophrenia represent an important dimension of psychopathology, and reflect the absence or diminution of normal behaviours and functions. They include deficiencies in emotional responsiveness, drive, and emotional and social engagement. Persistent negative symptoms are held to account for much of the long-term morbidity and poor functional outcome in patients with established schizophrenia, but if they prove resistant to antipsychotic medication there is a very limited evidence base regarding specific treatments. The aim of this double-blind, placebo-controlled trial is to establish the clinical and cost effectiveness of an SSRI antidepressant, citalopram, in the management of negative symptoms of schizophrenia over a year. The study sample will be adults with a diagnosis of schizophrenia, clinically stable for 3 months with a consistent antipsychotic regimen, and characterised by persistent negative symptoms to a criterion level of severity.

ELIGIBILITY:
Inclusion Criteria:

* An OPCRIT (Operational Criteria Checklist for Psychosis: 57) diagnosis of schizophrenia, schizophreniform, schizoaffective disorder or psychosis NOS as defined by DSM-IV.
* A negative subscale score of 20 or more on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS). At least three of the seven items on the negative symptom subscale should be rated 3 or more.
* Age 18-75 years, inclusive
* Clinically stable for the last 3 months with a consistent antipsychotic regimen.
* Competent and willing to provide written, informed consent.

Exclusion criteria:

* Any medical contraindications to an SSRI antidepressant.
* Currently receiving antidepressant or clinician wants to treat with an antidepressant;
* Taking any medications that risk interacting with citalopram
* Known congenital long QT syndrome, congestive heart failure, bradyarrhythmias
* QT limit above the upper limit of normal as determined by an electrocardiogram (ECG)
* Serum potassium and/or magnesium levels below the lower limits of normal
* Currently fulfil criteria for major depressive disorder; alcohol/substance hazardous use or dependence in past 3 months
* Treated with ECT in the last 8 weeks.
* Pregnant or planning to become pregnant
* Cognitive or language difficulties that would preclude subjects providing informed consent or compromise participation in study procedures.
* Lack of consent, as judged by the patient's psychiatrist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Barnes, MD, Principal Investigator — Imperial College London
Locations (14):
- United Kingdom (14):
  - Avon and Wiltshire mental health partnership, Bristol
  - Derbyshire healthcare NHS foundation trust, Derby
  - Lincolnshire partnership NHS foundation trust, Lincoln
  - West london Mental Health Trust, London
  - Camden and Islington NHS foundation trust, London
  - Central and North West London NHS foundation trust, London
  - Oxleas NHS foundation trust, London
  - South London and the Maudsley, London
  - Manchester health and social care trust, Manchester
  - Northumberland, Tyne and Wear NHS foundation trust, Newcastle
  - Oxfordshire and Buckinghamshire NHS foundation trust, Oxford
  - Sheffield social care foundation trust, Sheffield
  - Southern Health, Southampton
  - South Staffordshire and Shropshire NHS foundation trust, Stafford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barnes TR, Leeson VC, Paton C, Costelloe C, Simon J, Kiss N, Osborn D, Killaspy H, Craig TK, Lewis S, Keown P, Ismail S, Crawford M, Baldwin D, Lewis G, Geddes J, Kumar M, Pathak R, Taylor S. Antidepressant Controlled Trial For Negative Symptoms In Schizophrenia (ACTIONS): a double-blind, placebo-controlled, randomised clinical trial. Health Technol Assess. 2016 Apr;20(29):1-46. doi: 10.3310/hta20290. PMID 27094189

RESULTS

PARTICIPANT FLOW:
Groups:
- Citalopram: Citalopram: 20mg/day for the first 4 weeks, followed by the option to increase the dose to 40mg per day for the remainder of the study period.
- Placebo: Placebo: one placebo capsule for the first 4 weeks, followed by the option to increase the dose to two placebo capsules for the remainder of the study period.
Period: Overall Study
Arm/Group | Citalopram | Placebo
Started | 30 | 32
Completed | 19 | 23
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.02 (12.3) | 45.1 (12.3) | 44.11 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 26 | 22 | 48
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: PANSS Negative Symptom Score
Description: The Positive and Negative Syndrome Scale (PANSS) is a semi-structured interview to elicit symptom ratings for 30 symptoms of psychosis, each scored between 1-7. The negative symptoms subscale uses the individual items in the PANSS that Marder identified as negative symptom (blunted affect, emotional withdrawal, poor rapport, passive/ apathetic social withdrawal, motor retardation, active social avoidance and lack of spontaneity/flow of conversation). Scores on these individual items are summed to create the subscale score. The subscale has a range of 7 to 49, with higher scores indicate greater psychopathology
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 22 | 24
units on a scale | 21.5 (5) | 23 (6.2)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Equivalence — For the primary outcome, linear regression was used to determine mean difference between treatment groups. Differences between groups are presented as mean differences with associated 95% confidence interval (CI). Baseline values for variables were included as covariates in regression models and adjusted according to analysis of covariance. All analyses were conducted under the intention-to-treat principle; p = 0.36, Regression, Linear; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-4.91 to 1.80]

2. Primary Outcome: Heinrich's Quality of Life Scale Score
Description: The Heinrichs Quality of Life scale is a 21-item scale based on a semi-structured interview designed to assess deficit symptoms. Each items is scored from 0-6 and the total score is the sum of all item responses. The total score has a range of 0 to 126, with higher scores indicating better functioning.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 21 | 25
score on a scale | 52 (18.7) | 49.5 (20)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.68, Regression, Linear; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-9 to 14]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Citalopram | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 8/30 | 11/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=30) | Placebo (N=32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (20) | 5 (5)
Vomitting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 5 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No